CLINICAL TRIAL: NCT04461899
Title: Changes in Serum antimüllerian Hormone Levels in Patients 3 and 12 Months After Endometrioma Sclerotherapy
Acronym: ENDOPAL AMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL20_0002; 2020-A00118-31 (Other: ANSM)
Record Dates: First submitted 2020-06-29; First posted 2020-07-08 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Endometriosis Ovary
Keywords: endometrioma; sclerotherapy; ovarian reserve; antimüllerian hormone
MeSH Terms: conditions — Endometriosis | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sclerotherapy (Other): a sclerotherapy will be done in patients
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: Blood test — additional blood test will be done 3 and 12 months after endometrioma sclerotherapy.

SUMMARY:
Endometriosis affects 6-10% of women in childbearing age. It is a heterogeneous disease with three different forms: superficial endometriosis (peritoneal), ovarian endometrioma and deep pelvic endometriosis (subperitoneal).

Surgical management of endometriomas is justified in cases of significant clinical symptoms (like pain), especially in cases of resistance to medical treatment. Currently, laparoscopic cystectomy surgery is the recommended technique to treat ovarian endometrioma. However, it is now well demonstrated that this surgery significantly reduces the ovarian reserve.

Ethanol sclerotherapy is an alternative technique used to treat ovarian endometriomas. Several studies demonstrated the effectiveness and safety of this treatment, particularly in terms of preserving fertility. Regarding these reassuring data, many clinicians changed their practices and propose this technique as a first-line surgery.

Ovarian reserve comprises two elements: size of the primordial follicle stock and quality of the ovocytes. Antimüllerian hormone (AMH) has been shown to be the best marker of fertility.

The aim of this study is to observe changes in AMH levels after endometrioma sclerotherapy. This study is conducted in the Hospices Civils de Lyon, in 3 different sites.

ELIGIBILITY:
Inclusion Criteria:

* Patient in childbearing age from 18 to 42 years.
* Patient with uni- or bilateral endometrioma(s) without clinical and ultrasound criteria for ovarian carcinoma.
* A sclerotherapy is programmed.
* Patient affiliated to a social security scheme.
* Patient who gave consent for this research.

Exclusion Criteria:

* doubt about the endometriotic origin of the cyst
* suspect malignant ovarian disease.
* Pregnant or breastfeeding patient.
* Patient participating in other research with an exclusion period still in progress at the time of inclusion or those included in interventional research that interferes with the study protocol.
* Patient deprived of liberty by judicial or administrative decision.
* Patient (≥ 18 years old) under legal protection or unable to give consent.
* Patient does not speak French.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
AMH level | 3 months (+/-15 days) after endometrioma sclerotherapy

SECONDARY OUTCOMES:
AMH level | 12 months (+/-15 days) after endometrioma sclerotherapy
AMH level | 12 months after endometrioma sclerotherapy
  AMH level 3 and 12 months after endometrioma sclerotherapy
Endometrioma recurrence | 3 months (+/-15 days) after endometrioma sclerotherapy
  New endometrioma (≥ 2 cm) unilateral or bilateral, single or multiple
Endometrioma recurrence | 12 months (+/-15 days) after endometrioma sclerotherapy
  New endometrioma (≥ 2 cm) unilateral or bilateral, single or multiple

CONTACTS AND LOCATIONS:
Overall Officials: Gil DUBERNARD, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Hopital Femme Mère Enfant, Bron
  - Hopital de la Croix Rousse, Lyon
  - Hopital Lyon Sud, Pierre-Bénite